CLINICAL TRIAL: NCT05874479
Title: Reducing AIR Pollution Exposure to Lower Blood PRESSURE Among New York City Public Housing Residents
Acronym: AirPressureNYC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-00517
Record Dates: First submitted 2023-05-12; First posted 2023-05-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Blood Pressure
Keywords: self-measured morning home systolic blood pressure (AM H-SBP)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Portable Air Cleaner (PAC) (Experimental): Using a double-blind randomized process, active PACs (with HEPA filters inside) will be assembled and placed in the bedroom of study participants. Initiation of the PAC devices will occur at baseline on Day 0. After completion of enrollment, consent and the placement of PACs, electricity monitors, and PurpleAir monitoring, the PAC will be turned on. Participants will be instructed to keep the PACs on in bedrooms during the study duration, closing bedroom doors at night and during the day, when possible. The PAC will run for 24 hours on Day 0 of the study protocol before the 30-day treatment period begins. A kilowatt meter will be installed with the PAC to monitor electricity usage as a measure of adherence.
  Interventions: Device: Active PAC
- Sham PAC (Sham Comparator): Using a double-blind randomized process, sham PACs (with no filters inside) will be assembled and placed in the bedroom of study participants. Initiation of the PAC devices will occur at baseline on Day 0. After completion of enrollment, consent and the placement of PACs, electricity monitors, and PurpleAir monitoring, the PAC will be turned on. Participants will be instructed to keep PACs on in bedrooms during the study duration, closing bedroom doors at night and during the day, when possible. The PAC will run for 24 hours on Day 0 of the study protocol before the 30-day treatment period begins. A kilowatt meter will be installed with the PAC to monitor electricity usage as a measure of adherence.
  Interventions: Device: Sham PAC

INTERVENTIONS:
Device: Active PAC — The active PAC will contain HEPA filters inside the device.
  Arms: Active Portable Air Cleaner (PAC)
Device: Sham PAC — The sham PAC will contain no HEPA filters inside the device.
  Arms: Sham PAC

SUMMARY:
Fine particulate matter <2.5 µm (PM2.5) air pollution is the fifth leading risk factor for global mortality, with the largest portion of deaths due to cardiovascular disease (CVD). While several mechanisms are responsible, PM2.5-induced elevations in blood pressure (BP) may be relevant. Indoor portable air cleaners (PACs) are a novel approach to reduce exposure to PM2.5 and potentially lower blood pressure. The current study is being conducted to provide evidence that PACs reduce PM2.5 exposure and lower systolic blood pressure (SBP) in key patient populations.

ELIGIBILITY:
Inclusion Criteria:

* self-reported nonsmokers living in a nonsmoking household.
* adults living with hypertension (HTN) from NYC public housing.

Exclusion Criteria:

* History of major known arrhythmias (e.g. atrial flutter or fibrillation, ventricular tachycardia).
* Screening systolic BP ≥160 mm Hg or diastolic BP ≥100 mm Hg (i.e. severe hypertension by the 2017 ACC/AHA BP guideline).
* A change in drug regimen in the prior 2 weeks or a planned change in drug regimen during the first 30 days for those taking antihypertensive medication.
* Current smoking or living with an active smoker who smokes indoors
* Planned travel out of NYC for ≥2 weeks in next 6 months
* Incarcerated
* Pregnant
* Unable/unwilling to consent
* Established cardiovascular disease
* End-stage renal disease (chronic kidney disease stage IV or on dialysis)
* Barrier to technology use (e.g., visual or hearing impairment)
* Lung disease requiring oxygen
* Cancer receiving treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Average Self-Measured Morning Home Systolic Blood Pressure (AM H-SBP) over 30 Days | Up to Day 30
  Participants measure HBP every day between 6-9 am.

SECONDARY OUTCOMES:
Average Self-Measured Morning Home Systolic Blood Pressure (AM H-SBP) over 90 Days | Up to Day 90
  Participants measure HBP every day between 6-9 am.
Average Self-Measured Morning Home Systolic Blood Pressure (AM H-SBP) over 180 Days | Up to Day 180
  Participants measure HBP every day between 6-9 am.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Newman, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Jonathan.newman@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Jonathan.newman@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.